CLINICAL TRIAL: NCT05418621
Title: Does the Non-surgical Application of Enamel Matrix Derivative Reduce the Need of Periodontal Surgical Intervention in Subjects With Severe (Stage III) Periodontitis? A Randomized, Multicenter, Clinical Trial
Brief Title: Does the Non-surgical Application of Enamel Matrix Derivative Reduce the Need of Periodontal Surgical Intervention in Subjects With Severe (Stage III) Periodontitis?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, Full Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PERIO-EMD 3
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enamel Matrix Derivative application (Experimental): At the completion of the subgingival instrumentation, in all sites with PPD>6 mm, a solution of 24% EDTA, will be first applied with a sterile syringe with a thin blunt tip (25GX1/4"). The tip will be inserted in the gingival crevice and run apically on the instrumented root taking particular care in not penetrating the underlying soft tissues. The sites will be then copiously rinsed with both water-spray and by 5 sec passage of ultrasonic instrument's fine tip in the site with no contact to the root surface. After irrigation, a thorough drying of the site will be performed with an air-spray and a section of an orthodontic floss will be placed in all sites and left in the site for 1 minute at least. Thus, once Superfloss is removed in the test group, EMD (Emdogain FL®, Institute Straumann AG, Basel, Switzerland) will be applied with a dedicated syringe until overflowing from the pocket border, taking particular care in avoiding trauma to the tissues.
  Interventions: Drug: Enamel Matrix Derivative application
- Saline application (Placebo Comparator): At the completion of the subgingival instrumentation, in all sites with PPD>5 mm, a solution of 24% EDTA , will be first applied with a sterile syringe with a thin blunt tip (25GX1/4"). The tip will be inserted in the gingival crevice and run apically on the instrumented root taking particular care in not penetrating the underlying soft tissues. The sites will be then copiously rinsed with both water-spray and by 5 sec passage of ultrasonic instrument's fine tip in the site with no contact to the root surface. After irrigation, a thorough drying of the site will be performed with an air-spray and a section of an orthodontic floss will be placed in all sites and left in the site for 1 minute at least. Thus, once Superfloss is removed in the control group, a lavage of sterile saline will be applied with a syringe with a thin blunt tip until overflowing from the pocket border, taking particular care in avoiding trauma to the tissues.
  Interventions: Other: Saline application

INTERVENTIONS:
Drug: Enamel Matrix Derivative application — in the test group, EMD (Emdogain FL®, Institute Straumann AG, Basel, Switzerland) will be applied with a dedicated syringe until overflowing from the pocket border, taking particular care in avoiding trauma to the tissues.
  Arms: Enamel Matrix Derivative application
Other: Saline application — in the control group, a lavage of sterile saline will be applied with a syringe with a thin blunt tip until overflowing from the pocket border, taking particular care in avoiding trauma to the tissues.
  Arms: Saline application

SUMMARY:
Periodontal treatment relies on a sequential series of different phases that are usually incapsulated in three main phases: non-surgical treatment, surgical phase and, finally, supportive phase. Whilst, on the one hand not all patients may undergo surgical interventions, on the other hand non-surgical periodontal and supportive treatment are administered to all subjects affected by periodontitis. Both phases are constituted by closed, non-surgical, root instrumentation which is often carried out with similar techniques. Thus, non-surgical periodontal treatment (NSPT) is the one key stone of the treatment of periodontitis.

NSPT is very efficacious. A significant majority of the diseased sites are usually managed non-surgically (Graziani et al., 2017)). Moreover, bleeding on probing and symptoms are significantly decreased by NSPT. Importantly, NSPT is also capable to reduce systemic inflammation (Teeuw et al., 2014), improve glycaemic control (Sanz et al., 2018) and overall ameliorate oral health related quality of life (Graziani, Music, et al., 2019). Lastly, NSPT is cost effective as its costs are moderate and it may be performed by both dentists and hygienists.

Nevertheless, NSPT is often uncapable to solve an entire clinical case and surgical treatment is advocated as in fact the complete closure of the pockets ranges from 57 to 75% according to a follow-up of 3⁄4 months or 6/8 respectively (Solini et al., 2019). Periodontal surgery is also effective, but it is nonetheless a surgical intervention which cannot be defined as deprived of side effects (Graziani et al., 2018).

Thus, in order to improve the outcome of NSPT numerous adjunctive treatment modalities have been advocated (Braun et al., 2008; Graziani et al., 2017; Haffajee et al., 2003). Yet the objective of reducing the need for surgery has been rarely evaluated.

Recently, our group ran a trial in which enamel matrix derivatives (EMD) has been applied as non-surgical adjunct. The findings highlighted that EMD application lowers systemic inflammation, increases blood clot stability and, locally, reduces of the need for surgery by 32% compared to the control group without EMD.

Thus, a multicentre responding to the following questions:

* Flapless application of EMD reduce the need for periodontal surgery?
* Are the results stable over time?
* Can the results be generalized among different clinicians? EMD is a resorbable, implantable material and supports periodontal regeneration, which takes place over more than a year. It consists of hydrophobic enamel matrix proteins extracted from developing embryonal enamel of porcine origin in a propylene glycol alginate carrier.

The gel has a suitable viscosity to facilitate application directly onto root surfaces exposed during periodontal surgery. Once applied onto an exposed root surface the protein self assembles into an insoluble three-dimensional matrix and creates a suitable environment for selective periodontal cell migration and attachment, which re-establishes lost tooth supporting tissues. Subsequent to formation of new attachment, alveolar bone can also be regenerated due to the osteogenic capacity of the restored periodontal ligament. EMD is degraded by enzymatic processes of normal wound healing.

ELIGIBILITY:
Inclusion Criteria

* Accept the form of the study and signs a declaration of informed consent; understand and are willing, able and likely to comply with all study procedures and restrictions.
* Systemically healthy (according to exclusion criteria 4) participants of either genders who are attending a periodontal centre for periodontal care.
* Aged 18 or over.
* Presenting at least 20 teeth (excluded wisdom teeth).
* Being affected by generalized Periodontitis (stage III) irrespectively of the grade (Tonetti et al., 2018) i.e. presenting at least 5 mm of clinical atattachment loss at the interdental areas, radiographic bone resorption of more than 30% of the root length extending to at least the middle portion of the root, less than 5 teeth lost for periodontal reason, presenting characteristics for complexity (intrabony defects, furcation defects, moderate ridge defects)
* Bleeding on probing on at least 30% of the sites and a minimum of 4 teeth with at least one site with PPD ≥6mm

Exclusion Criteria:

* Persons incapable of responding to the questions.
* An employee of the sponsor, employee of the general dental practice, and/or a family relative of the employees mentioned above.
* Women known to be pregnant or lactating (a specific declaration form will be signed by the patient, stating the non-pregnant or lactating status).
* Persons suffering of pathologies known to affect the outcome of periodontal therapy (i.e. diabetes, osteoporosis, immunosuppression).
* Persons undergoing therapy which will may complicate adherence to protocol or showing an impact on periodontal outcome (i.e. chemotherapy and immunosuppressive treatments).
* Persons who require antibiotic coverage (following infectious endocarditis, using prosthetic cardiac valves, other pathologies).
* Persons undergoing pharmacological treatment associated with gingival hypertropia development (phenytoin, phenobarbital, lamotrigine, vigabatrin, ethosuximide, topiramate, primidone, nifedipine, amlodipine, verapamil, cyclosporine).

Persons with implant-supported restorations affected by peri-implantitis (as defined by the 2017 Classification, i.e. presence of bleeding and/or suppuration on gentle probing, probing depths of ≥6 mm, bone levels ≥3 mm apical of the most coronal portion of the intraosseous part of the implant).

* Smokers declaring to smoke more than 20 cigarettes per day.
* Persons with Body Mass Index above 29(obese subjects).
* Anyone who in the investigators' opinion is not suitable to take part in the study.
* Allergy/idiosyncrasy to anaesthesia or components of the device object of the study.
* Previous periodontal subgingival instrumentation within the previous 12 months.
* Antibiotics intake in the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Resolved cases | 3, 6 and 12 months after treatment
  inter-group differences in % of cases, patient-level analysis, with complete absence of sites with Probing Pocket Depth (PPD) >=6mm

SECONDARY OUTCOMES:
number of sites with PPD>=6mm | 3, 6 and 12 months after treatment
  Intra-group and intergroup changes in % and number of sites with PPD>=6mm. The Probing Pocket Depth (PPD) will be measured as the distance between the gingival margin and the deepest part of the gingival pocket measured through a University of North Carolina -15 periodontal probe (UNC-15) (Hu-Friedy, USA). PPD will be evaluated at 6 sites on each tooth: disto-buccal, buccal, mesio-buccal, disto-lingual, lingual, mesio-lingual. Each measure will be rounded to the nearest millimetre probe.
changes in Full Mouth Plaque Score (FMPS) | 3, 6 and 12 months after treatment
  intragroup and intergroup change in Full Mouth Plaque Score. The Full Mouth Plaque Score (FMPS) will be measured as the presence or absence of plaque on each tooth surface will be assessed. The bacterial deposits are stained with a plaque-disclosing solution (erythrosine). Areas adjacent to the gingival margins that exhibit an intense staining that can be easily removed with the edge of the probe will be dotted as having plaque. The presence of plaque will be evaluated as 1, while the absence as 0 on 6 areas per tooth (disto-buccal, buccal, mesio- buccal, disto-lingual, lingual, mesio-lingual). A dedicated diagram (see attached medical records, chapter 16) will allow to draw the overall plaque accumulation and mean plaque score will be indicated in percentage (% of sites found positive for the presence of plaque on the total of 6 sites per tooth (O'Leary et al., 1972).
changes in Full Mouth Bleeding Score (FMBS) | 3, 6 and 12 months after treatment
  intragroup and intergroup change in Full Mouth Bleeding Score. The Full Mouth Bleeding Score (FMBS) will be measured dichotomously after periodontal probing. It will be considered positive when the bleeding occurs after the retraction of the probe (approximate time for evaluation 30 seconds after probe insertion). It will be considered negative when there is no bleeding. The mean bleeding score is indicated in percentage (% of sites detected positive for bleeding on the total 6 sites per tooth )(Ainamo & Bay, 1975).
mean values of PPD | 3, 6 and 12 months after treatment
  Intra-group and intergroup changes in terms of full mouth mean values of PPD. The Probing Pocket Depth (PPD) will be measured as the distance between the gingival margin and the deepest part of the gingival pocket measured through a University of North Carolina -15 periodontal probe (UNC-15) (Hu-Friedy, USA). PPD will be evaluated at 6 sites on each tooth: disto-buccal, buccal, mesio-buccal, disto-lingual, lingual, mesio-lingual. Each measure will be rounded to the nearest millimetre probe.
mean values of recession (REC) | 3, 6 and 12 months after treatment
  Intra-group and intergroup changes in terms of full mouth mean values of REC. The Recession (Rec) will be measured as the distance in mm from the cement-enamel junction (CEJ) to the gingival margin measured through UNC- 15. In the event that CEJ would not be available, one of the following clinical landmarks will be used: crown margin, restored margin, occlusal point.
mean values Clinical Attachment Level (CAL) | 3, 6 and 12 months after treatment
  Intra-group and intergroup changes in terms of full mouth mean values of CAL. CAL will be calculated as the sum of PPD and REC.
Furcation involvement | 3, 6 and 12 months after treatment
  Intragroup and intergroup changes in terms of furcations degree. Furcation (FI): furcation involvements will be classified according to horizontal probing with Naber's probe in degree I when the probe can enter the orifice of the furcation, degree II when the probe can enter the furcation freely without passing it completely. Class III will be scored when the tip of the Nabers probe will see appearing through the opposite cervice, i.e. "through-and.through" furcation in both mandibular and maxillary molar (Hamp et al., 1975).
Dentine sensitivity (Schiff test) | 3, 6 and 12 months after treatment
  Intra-group and intergroup changes of dentine hypersensitivity as measured with the Schiff test. Schiff test: dentine sensitivity will be assessed trough the study timepoints as reported further using a validated a well described test as the Schiff test (Schiff et al., 1994). The Schiff test is a non-invasive and safety test that consist in spraying air on the tooth and collecting the reaction of the patient in a liker type scale as follows:
  * 0 Subject does not respond to air stimulus;
  * 1 Subject responds to air stimulus but does not request discontinuation of stimulus;
  * 2 Subject responds to air stimulus and requests discontinuation of stimulus;
  * 3 Subject responds to air stimulus, considers stimulus to be painful and requests discontinuation of stimulus.
Oral Health Impact profile 14 | 3, 6 and 12 months after treatment
  Oral Health Index Profile-14 (OHIP-14): a validated questionnaire of 14 question aiming at assessing statements grouped in 7 conceptual subscales: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. It allows an evaluation of the OHRQoL (Slade, 1997). The higher the score, the higher the impact of periodontitis on the patients quality of life
Attention Network Task | 3, 6 and 12 months after treatment
  Attention Network Task (ANT; Fan et al., 2002): a task designed to test three attentional networks: alerting, orienting, and executive control.The higher the score, the higher the cognitive abilities.
Corsi block-tapping test | 3, 6 and 12 months after treatment
  Corsi block-tapping test (CBTT; Orsini et al., 1987): a task to assess visuo-spatial short-term memory. The higher the score the better the cognitive ability
Tower of London | 3, 6 and 12 months after treatment
  Tower of London (ToL; Shallice, 1982): a task designed to evaluate problem-solving and planning capabilities.The higher the score the better the cognitive abilities
Sickness Questionnaire | 3, 6 and 12 months after treatment
  Sickness Questionnaire ( SicknessQ ; Andreasson et al., 2018): a brief instrument, composed of 10 items, aimed to assess perceived sickness behaviour. The higher the score the higher the perceived thickness
Depression Anxiety Stress Scale | 3, 6 and 12 months after treatment
  Depression Anxiety Stress Scale - 21 (DASS-21; Lovibond & Lovibond, 1995): self - report questionnaire designed to assess the symptoms of depression, anxiety and stress. The higher the score the higher the symptoms of depression, anxiety and stress.
State-Trait Anxiety Inventory_ Form | 3, 6 and 12 months after treatment
  State-Trait Anxiety Inventory_ Form Y2 ( STAI_Y2; Spielberger, 1983): self - report questionnaire aimed to investigate trait anxiety that refers to relatively stable individual differences in anxiety proneness, that is, to differences between people in the tendency to perceive stressful situation as dangerous or threatening. The higher the score the higher the tendency os being prone to anxiety.
State-Trait Anxiety Inventory_ Form Y1 | 3, 6 and 12 months after treatment
  State-Trait Anxiety Inventory_ Form Y1 ( STAI_Y1; Spielberger, 1983): self - report questionnaire aimed to investigate trait anxiety that refers to a palpable reaction or process taking place at a given time and level of intensity. The higher the score the higher the trait of anxiety assessed.
Profile Mood State | 3, 6 and 12 months after treatment
  Profile of Mood State (POMS; Grove, Robert & Prapavessis, 2016): self - report questionnaire aimed to investigate different mood states like.: tension, depression, anger, fatigue, confusion and vigour.
Sleep quality | 3, 6 and 12 months after treatment
  Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 1989): self-assessment scale that provides a reliable, valid and standardized measure of sleep quality. The higher the score the better the sleep quality
The Insomnia Severity Index | 3, 6 and 12 months after treatment
  The Insomnia Severity Index (ISI; Morin, 1993): is a self-report questionnaire designed to assess the nature, severity and daytime impact of insomnia. The higher the score the higher the severity of insomnia.
Epworth Sleepiness Scale | 3, 6 and 12 months after treatment
  Epworth Sleepiness Scale (ESS; Johns, 1991): is a self-assessment tool consisting of 8 items that investigate the general level of daytime sleepiness or the propensity to sleep during different situations of daily life. The higher the score the higher the daily sleepiness.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University Hospital of Pisa, Pisa
  - Azienda Ospedaliero Universitaria Pisana, Pisa

IPD SHARING:
Plan to Share IPD: Undecided